CLINICAL TRIAL: NCT00807170
Title: A Phase I Study of ZD6474 (Vandetanib) Concurrent With Whole Brain Radiotherapy for the Treatment of Brain Metastases in Patients With Non-small Cell Lung Cancer (NSCLC)
Brief Title: Investigate the Maximum Tolerated Dose of Vandetanib and Concurrent Whole Brain Radiotherapy (WBRT) in Patients With Non-small Cell Lung Cancer (NSCLC) and Brain Metastases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Very slow recruitment
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4200C00085; EUDRACT Number 2008-005556-24
Record Dates: First submitted 2008-12-09; First posted 2008-12-11 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Non-small Cell Lung Cancer (NSCLC); Whole Brain Radiotherapy; metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ZACTIMA TM (Experimental)
  Interventions: Drug: ZD6474 (Vandetanib); Radiation: Whole Brain Radiotherapy (WBRT); Drug: ZD6474

INTERVENTIONS:
Drug: ZD6474 (Vandetanib) — 100 mg as a once daily oral dose, 21 days
  Other Names: ZACTIMA TM
Radiation: Whole Brain Radiotherapy (WBRT)
Drug: ZD6474 — 200 mg as a once daily oral dose, 21 days
  Other Names: ZACTIMA TM
Drug: ZD6474 — 300 mg as a once daily oral dose, 21 days
  Other Names: ZACTIMA TM

SUMMARY:
A clinical study to investigate the maximum tolerated dose of Vandetanib and concurrent WBRT in patients with NSCLC and brain metastases. All patients will receive WBRT, 10 fractions of 3 Gy. Patients will start 7 days prior to start of radiation treatment with Vandetanib. Total treatment time with Vandetanib is 3 weeks (21 days). Patients will have the opportunity to continue Vandetanib until progression at a dose of 300 mg. This multi-centre study will be conducted in a minimum of 9 patients and a maximum of 18 patients at 3 sites.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged above 18 years with histologically or cytologically confirmed NSCLC and contrast-enhanced CT scan or Gadolinium-enhanced MRI confirmed brain metastases who have a performance status of 0 to 2
* No previous radiotherapy, surgery or chemotherapy for brain metastases
* Patients should not have any unstable systemic disease

Exclusion Criteria:

* Serious abnormal laboratory values
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol
* Clinically significant cardiovascular event (e.g. myocardial infarction, superior vena cava syndrome (SVC), New York Heart Association (NYHA) classification of heart disease >2 within 3 months before entry; or presence of cardiac disease that, in the
* Previous randomization of treatment in the present study and/ or current participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To investigate the maximum tolerated dose of Vandetanib and concurrent WBRT in patients with NSCLC and brain metastases | All evaluable patients (all registered patients who receive at least opne dose of study medication) who have completed week 9 study period

SECONDARY OUTCOMES:
To investigate the time to clinical and radiological progression of brain metastases | Until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- Netherlands (3):
  - Research site, Amsterdam
  - Research site, Groningen
  - Research site, Maastricht